CLINICAL TRIAL: NCT00413010
Title: An 8-Week, Double-Blind, Placebo-Controlled, Phase 3 Trial of Pregabalin (150-600 mg/Day) in the Adjunctive Treatment of Patients With Generalized Anxiety Disorder (GAD) Who Have Not Optimally Responded to Existing Therapies(GAD)
Brief Title: Pregabalin in the Treatment of Patients With Generalized Anxiety Disorder (GAD).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081103
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2009-12

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo
- Arm 1 (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — pregabalin 150-600 mg/day flexibly dosed for the first 6 weeks and fixed dosed for the last 2 weeks of total 8 weeks of double blind study period, + concurrent GAD treatment from the open-label study period
  Other Names: Lyrica
  Arms: Arm 1
Drug: placebo — placebo + concurrent GAD treatment from the open-label study period
  Arms: Arm 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy of pregabalin as compared to placebo in the treatment of patients with general anxiety disorder (GAD). Efficacy will be measured by the improvement in the total Hamilton Anxiety Rating Scale (HAM-A) scores from baseline observed following 8 weeks of double-blind treatment or at earlier termination during the double-blind treatment phase and analyzed using a mixed linear model for repeated measures.

DETAILED DESCRIPTION:
Further enrollment in this study was stopped on January 28, 2008 based on the recommendation of an independent data monitoring committee. The recommendation to stop the study was not based on any safety findings.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects with primary DSM-IV diagnosis of GAD, as confirmed by the MINI structured interview.
* Historical failure to respond optimally to a GAD treatment

Exclusion Criteria:

* Current primary DSM-IV (Diagnostic and Statistical Manual of Mental Disorders 4th edition) diagnosis of major depressive disorder with or without seasonal pattern, dysthmic disorder, depressive disorder NOS (not otherwise specified), social phobia, panic disorder with or without agoraphobia, post traumatic stress disorder, dissociative disorder, borderline personality disorder, obsessive-compulsive disorder, antisocial personality disorder, as defined in the DSM-IV TR (Diagnostic and Statistical Manual of Mental Disorders 4th edition, Text Revision).
* Past and/or current DSM-IV diagnosis of schizophrenia, schizoaffective disorder, other psychotic disorders, bipolar disorders (I or II), factitious disorder or cognitive disorder (including delirium, dementia, and amnestic disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (31):
  - Pfizer Investigational Site, Arcadia, California
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, Sherman Oaks, California
  - Pfizer Investigational Site, Norwich, Connecticut
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Fort Walton Beach, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Saint Charles, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Waukesha, Wisconsin
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Litoměřice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 8 - Bohnice
- Estonia (3):
  - Pfizer Investigational Site, Viljandi, Viljandi Mk.
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Finland (3):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Joensuu
  - Pfizer Investigational Site, Kuopio
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Pécs
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
- Serbia (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Kragujevac
- Ukraine (5):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Luhansk
  - Pfizer Investigational Site, Lviv

REFERENCES:
- [Derived] Rickels K, Shiovitz TM, Ramey TS, Weaver JJ, Knapp LE, Miceli JJ. Adjunctive therapy with pregabalin in generalized anxiety disorder patients with partial response to SSRI or SNRI treatment. Int Clin Psychopharmacol. 2012 May;27(3):142-50. doi: 10.1097/YIC.0b013e328350b133. PMID 22302014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 55 centers in 8 countries (United States, Russian Federation, Czech Republic, Ukraine, Serbia, Hungary, Finland, and Estonia).
Pre-assignment Details: After a screening phase (Period 1), subjects entered an 8-week open-label treatment optimzation phase (Period 2). Only those subjects who partially responded to background Generalized Anxiety Disorder (GAD) treatment (escitalopram, paroxetine, or venlafaxine XR) and met all inclusion/exclusion criteria were eligible for randomization (Period 3).
Groups:
- Pregabalin: Pregabalin doses of 150 milligrams (mg)/day, 300 mg/day, 450 mg/day, and 600 mg/day was administered orally, twice daily (BID), with or without food, during the double-blind phase. Flexible dosing of pregabalin was allowed during the first 6 weeks; fixed dosing was required for the last 2 weeks of this period.Subjects were required to remain on a stable dose of their concurrent Generalized Anxiety Disorder (GAD) treatment (ie, escitalopram, paroxetine, or venlafaxine XR).
- Placebo: Placebo was administrated orally, twice daily (BID) with or without food, during the double-blind phase. Subjects were required to remain on a stable dose of their concurrent GAD treatment (ie, escitalopram, paroxetine, or venlafaxine XR).
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 180 | 176
Completed | 108 | 113
Not Completed | 72 | 63
Not completed — Adverse Event | 8 | 4
Not completed — Laboratory abnormality | 0 | 2
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Due to termination of the study | 54 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 180 | 176 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.5) | 43.5 (12.5) | 43.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 115 | 244
  Male | 51 | 61 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Anxiety Rating Scale (HAM-A) Total Scores
Description: Change from baseline: average across visit weeks using mixed model. HAM-A=clinician-rated interview measuring presence of anxiety-related symptoms in 14 areas including anxiety, tension, depressed mood, palpitations, breathing difficulties, sleep disturbances, & restlessness. Total score ranges from 0 to 56; higher score indicates greater anxiety.
Time Frame: Baseline, 8 weeks
Population: Intent-to-Treat (ITT) population included all randomized subjects who had received at least 1 dose of the double-blind treatment. All efficacy analyses included the ITT subjects who had a Baseline and a post-Baseline assessment of the respective efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
score on scale | -7.6 (0.35) | -6.4 (0.36)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Null hypothesis: no difference between Pregabalin (150-600 mg/day) BID and Placebo BID treatment groups. An initial sample size of 173 subjects per double-blind treatment group was calculated to provide at least 90% power to detect an effect size (ie, difference in the true means between 2 treatment groups/standard deviation) of 0.36 for the HAM-A total score change from Baseline using a 2-sided nominal significance level of 4.9%; Test type: Superiority or Other; Mixed Models Analysis; Adjusted for treatment, pooled center baseline, HAM-A total score,time,and treatment-by time; Mean Difference (Final Values) = -1.2, 95% CI [-2.16 to -0.26], Standard Error of Mean 0.48 — Since an interim analysis was conducted and the sample size was larger than the targeted 173 subjects per group, a critical t-value adjustment was 1.977, yielding an adjusted 95% CI shown above

2. Secondary Outcome: Change in HAM-A Total Score at Weekly Visits
Description: Change: score at each study week minus score at baseline. HAM-A, a clinician-rated interview, measures presence of anxiety-related symptoms in 14 areas including anxiety, tension, depressed mood, palpitations, breathing difficulties, sleep disturbances, & restlessness. Total score ranges from 0 to 56; higher score indicates greater anxiety.
Time Frame: Baseline, Weeks 1 through Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
score on scale
  Week 1 (n=164;n=169) | -4.4 (0.37) | -3.1 (0.37)
  Week 2 (n=166;n=163) | -6.3 (0.43) | -5.2 (0.43)
  Week 3 (n=157;n=160) | -7.0 (0.45) | -5.5 (0.45)
  Week 4 (n=153;n=150) | -8.3 (0.46) | -7.0 (0.47)
  Week 5 (n=135;n=130) | -8.4 (0.49) | -7.6 (0.49)
  Week 6 (n=122;n=125) | -9.2 (0.49) | -8.0 (0.49)
  Week 8 (n=126;n=127) | -9.3 (0.56) | -8.0 (0.56)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Treatment (tx) adjusted, pooled center baseline HAM-A total score,time,and tx-by time. Degrees of freedom adjusted using Satterthwaite approximation; Mean Difference (Final Values) = -1.33, 95% CI [-2.3 to -0.4], Standard Error of Mean 0.49 — Difference reflects pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Median Difference (Final Values) = -1.04, 95% CI [-2.2 to 0.1], Standard Error of Mean 0.59 — Difference reflects pregabalin minus placebo
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.45, 95% CI [-2.7 to -0.2], Standard Error of Mean 0.62 — Difference reflects pregabalin minus placebo
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.33, 95% CI [-2.6 to -0.1], Standard Error of Mean 0.64 — Difference reflects pregabalin minus placebo
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.78, 95% CI [-2.1 to 0.5], Standard Error of Mean 0.68 — Difference reflects pregabalin minus placebo
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.22, 95% CI [-2.5 to 0.1], Standard Error of Mean 0.67 — Difference reflects pregabalin minus placebo
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.35, 95% CI [-2.9 to 0.2], Standard Error of Mean 0.77 — Difference reflects pregabalin minus placebo

3. Secondary Outcome: Number of Responders Using Hamilton Anxiety Rating Scale (HAM-A)
Description: Responders = YES if subjects achieved a >= 50% decrease in HAM-A total score from Baseline to respective study week. HAM-A is a clinician-rated interview measuring the presence of anxiety-related symptoms in 14 areas. Total score ranges from 0 to 56; higher score indicates greater anxiety.
Time Frame: Weeks 1 through Week 8
Population: Intent-to-Treat (ITT) population included all randomized subjects who had received at least 1 dose of the double-blind treatment, and had a baseline and post-baseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
participants
  Week 1 Responder: Yes | 21 | 8
  Week 1 Responder: No | 143 | 161
  Week 2 Responder: Yes | 39 | 26
  Week 2 Responder: No | 127 | 137
  Week 3 Responder: Yes | 51 | 23
  Week 3 Responder: No | 106 | 137
  Week 4 Responder: Yes | 64 | 46
  Week 4 Responder: No | 89 | 104
  Week 5 Responder: Yes | 58 | 46
  Week 5 Responder: No | 77 | 84
  Week 6 Responder: Yes | 57 | 48
  Week 6 Responder: No | 65 | 77
  Week 8 Responder: Yes | 63 | 47
  Week 8 Responder: No | 63 | 80
  Week 8 (LOCF) Responder: Yes | 84 | 62
  Week 8 (LOCF) Responder: No | 93 | 114
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; Regression, Logistic — P-value less that the nominal 0.05 level is suggestive of a treatment difference; P-value corresponds to Wald's Chi square test; Based on fitting a logistic regression on the HAM-A responders at each week with treatment and center in the model; Odds Ratio (OR) = 3.35, 95% CI [1.37 to 8.24] — The odds ratio represented the odds of demonstrating an improvement comparing pregabalin versus placebo. Odds of being a responder (yes) for pregabalin relative to the odds of being a responder for placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Test type: Superiority or Other; Regression, Logistic — P-value less than the nominal 0.05 level is suggestive of a treatment difference; P-value corresponds to Wald's Chi square test; Based on fitting a logistic regression on the HAM-A responsers at each each with treatment and center in the model; Odds Ratio (OR) = 1.61, 95% CI [0.90 to 2.87] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the HAM-A responsers at each each with treatment and center in the model; Odds Ratio (OR) = 3.15, 95% CI [1.76 to 5.66] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the HAM-A responsers at each each with treatment and center in the model; Odds Ratio (OR) = 1.80, 95% CI [1.06 to 3.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the HAM-A responsers at each each with treatment and center in the model; Odds Ratio (OR) = 1.57, 95% CI [0.90 to 2.73] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the HAM-A responsers at each each with treatment and center in the model; Odds Ratio (OR) = 1.52, 95% CI [0.86 to 2.66] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the HAM-A responsers at each each with treatment and center in the model; Odds Ratio (OR) = 1.86, 95% CI [1.08 to 3.22] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8 (last observation carried forward, LOCF); Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the HAM-A responders at Week 8 (LOCF) with treatment and center in the model; Odds Ratio (OR) = 1.77, 95% CI [1.12 to 2.79] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Subjects in Remission Using Hamilton Anxiety Rating Scale (HAM-A) Total Score
Description: Participant in remission defined as HAM-A total score of <= 7. HAM-A=clinician-rated interview measuring presence of anxiety-related symptoms in 14 areas including anxiety, tension, depressed mood, palpitations, breathing difficulties, sleep disturbances, & restlessness. Total score ranges 0 - 56; higher score indicates greater anxiety.
Time Frame: Week 1 through Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
participants
  Week 1 Remission: Yes | 12 | 5
  Week 1 Remission: No | 152 | 164
  Week 2 Remission: Yes | 22 | 15
  Week 2 Remission: No | 144 | 148
  Week 3 Remission: Yes | 32 | 18
  Week 3 Remission: No | 125 | 142
  Week 4 Remission: Yes | 43 | 29
  Week 4 Remission: No | 110 | 121
  Week 5 Remission: Yes | 39 | 30
  Week 5 Remission: No | 96 | 100
  Week 6 Remission: Yes | 37 | 32
  Week 6 Remission: No | 85 | 93
  Week 8 Remission: Yes | 40 | 31
  Week 8 Remission: No | 86 | 96
  Week 8 (LOCF) Remission: Yes | 55 | 42
  Week 8 (LOCF) Remission: No | 122 | 134
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 2.88, 95% CI [0.94 to 8.80] — The odds ratio represented the odds of demonstrating an improvement comparing pregabalin versus placebo. Odds of being a remitter (yes) for pregabalin relative to the odds of being a remitter for placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 1.49, 95% CI [0.72 to 3.06] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 2.08, 95% CI [1.09 to 3.97] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 1.80, 95% CI [0.99 to 3.28] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 1.53, 95% CI [0.82 to 2.85] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 1.33, 95% CI [0.71 to 2.48] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on fitting a logistic regression on the HAM-A remission at Week 8 with treatment and center in the model; Odds Ratio (OR) = 1.55, 95% CI [0.85 to 2.83] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8 Last Observation Carried Foward (LOCF); Test type: Superiority or Other; Regression, Logistic; Based on fitting a logistic regression on the HAM-A responders at Week 8 (LOCF) with treatment and center in the model; Odds Ratio (OR) = 1.53, 95% CI [0.92 to 2.53] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Time to Onset of Sustained Hamilton Anxiety Rating Scale (HAM-A) Improvement
Description: Time to sustained improvement was defined as time to 50% or greater reduction in HAM-A total score from Baseline, which was sustained for the remainder of the study. HAM-A is a clinician-rated interview measuring the presence of anxiety-related symptoms in 14 areas. Total score ranges from 0 to 56; a higher score indicates greater anxiety.
Time Frame: Week 8
Population: Intent-to-Treat (ITT) population included all randomized subjects who had received at least 1 dose of the double-blind treatment, and had a baseline and post-baseline efficacy assessment. CI for placebo patients was not estimable.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 0
days | 57 [43.0 to 61.0] |
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Kaplan Meier product limit estimate for calculating median time in days to onset sustained HAM-A Improvement; Test type: Superiority or Other; p = 0.0137, Log Rank — P-value corresponds to the 2-sided log-rank test; 2-sided log-rank test

6. Secondary Outcome: Number of Responders Using Clinical Global Impression of Improvement (CGI-I) Score
Description: Responders = YES using CGI-I if score indicated much improved or very much improved at the last study week. CGI-I is a clinician-rated instrument that measures change in subject's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 1 through Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
participants
  Week 1: Yes | 62 | 49
  Week 1: No | 101 | 120
  Week 2: Yes | 94 | 74
  Week 2: No | 72 | 89
  Week 3: Yes | 93 | 76
  Week 3: No | 62 | 86
  Week 4: Yes | 97 | 88
  Week 4: No | 55 | 61
  Week 5: Yes | 89 | 81
  Week 5: No | 45 | 50
  Week 6: Yes | 83 | 76
  Week 6: No | 38 | 49
  Week 8: Yes | 80 | 82
  Week 8: No | 43 | 45
  Week 8 (LOCF): Yes | 113 | 110
  Week 8 (LOCF): No | 61 | 66
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression on the CGI-I responders at Week 8 with treatment and center in the model; Odds Ratio (OR) = 1.54, 95% CI [0.96 to 2.47] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.58, 95% CI [1.01 to 2.47] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.75, 95% CI [1.09 to 2.82] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.26, 95% CI [0.77 to 2.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.24, 95% CI [0.72 to 2.11] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; Regression, Logistic; P-value less than the nominal 0.05 level is suggestive of a treatment difference; P-value corresponds to Wald's Chi square test; Odds Ratio (OR) = 1.45, 95% CI [0.84 to 2.50] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.06, 95% CI [0.61 to 1.84] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8 (LOCF) Last Observation Carried Forward; Test type: Superiority or Other; Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Odds Ratio (OR) = 1.12, 95% CI [0.71 to 1.76] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Clinical Global Impression of Severity (CGI-S) Score
Description: CGI-S is a clinician-rated instrument measuring the severity of a subject's symptoms on a 7-point categorical scale. Scores range from 1 (not at all ill) to 7 (among the most extremely ill patients). Higher score indicates that the subject is more ill.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
participants
  Normal, not ill at all | 28 | 18
  Borderline, mentally ill | 49 | 37
  Mildly ill | 49 | 63
  Moderately ill | 46 | 48
  Markedly ill | 2 | 8
  Severely ill | 2 | 1
  Among the most extremely ill | 0 | 0
  Not assessed | 0 | 1
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 8 Last Observation Carried Forward (LOCF); Test type: Superiority or Other; Cumulative Logit Model — [p-value comment as in outcome 3, analysis 2]; Based on fitting a logistic regression model for ordinal response of CGI-S scores at Week 8 (LOCF) with treatment and center in the model; Odds Ratio (OR) = 1.56, 95% CI [1.07 to 2.30] — The odds ratio represented the odds of demonstrating an improvement comparing pregabalin versus placebo. The odds of having an increasingly better response for pregabalin relative to the odds of having an increasingly better response for placebo

8. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) Total Score
Description: Change: score at each study week minus score at baseline. HAM-D, clinician-rated interview, measures presence of depressive symptoms in 17 areas (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, & weight loss). Total score ranges from 0 to 52; higher scores indicate more depression.
Time Frame: Weeks 1 through Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 177 | 176
score on scale
  Week 1 n=165,168 | -2.1 (0.28) | -1.3 (0.28)
  Week 2 n=165,164 | -3.1 (0.30) | -2.4 (0.31)
  Week 3 n=156,160 | -3.5 (0.32) | -2.8 (0.32)
  Week 4 n=153, 149 | -4.7 (0.29) | -3.3 (0.29)
  Week 5 n=135, 130 | -4.3 (0.33) | -3.9 (0.34)
  Week 6 n=122, 125 | -4.7 (0.33) | -3.8 (0.33)
  Week 8 n= 126, 127 | -4.8 (0.40) | -3.8 (0.40)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; ANCOVA; Repeated analysis of covariance heterogeneous auto-regressive w/ tx center wk & tx by wk fixed effects; Baseline HAM-D total score covariate in model; Mean Difference (Final Values) = -0.8, 95% CI [-1.5 to 0.0] — Difference is pregabalin minus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI [-1.5 to 0.2] — Difference is pregabalin minus placebo
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-1.6 to 0.1] — Difference is pregabalin minus placebo
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI [-2.1 to -0.6] — Difference is pregabalin minus placebo
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-1.3 to 0.5] — Difference is pregabalin minus placebo
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI [-1.8 to 0.0] — Difference is pregabalin minus placebo
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 8; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI [-2.1 to 0.1] — Difference is pregabalin minus placebo

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 3
Other Adverse Events (participants affected / at risk) | 81 | 59
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pregabalin | Placebo
Cardiac failure congestive (Cardiac disorders) | 1/180 | 0/176
Cellulitis (Infections and infestations) | 1/180 | 0/176
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1/180 | 0/176
Depression (Psychiatric disorders) | 0/180 | 1/176
Abdominal pain upper (Gastrointestinal disorders) | 0/180 | 1/176
Lower limb fracture (Injury, poisoning and procedural complications) | 0/180 | 1/176
Fall (Injury, poisoning and procedural complications) | 0/180 | 1/176
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin | Placebo
Vision blurred (Eye disorders) | 8/180 | 2/176
Constipation (Gastrointestinal disorders) | 5/180 | 3/176
Diarrhea (Gastrointestinal disorders) | 7/180 | 7/176
Dry mouth (Gastrointestinal disorders) | 4/180 | 2/176
Dyspepsia (Gastrointestinal disorders) | 6/180 | 1/176
Flatulence (Gastrointestinal disorders) | 4/180 | 0/176
Nausea (Gastrointestinal disorders) | 13/180 | 8/176
Vomiting (Gastrointestinal disorders) | 2/180 | 4/176
Fatigue (General disorders) | 7/180 | 5/176
Nasopharyngitis (Infections and infestations) | 5/180 | 6/176
Upper respiratory tract infection (Infections and infestations) | 3/180 | 6/176
Weight increased (Investigations) | 4/180 | 0/176
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/180 | 1/176
Dizziness (Nervous system disorders) | 21/180 | 10/176
Headache (Nervous system disorders) | 17/180 | 7/176
Paraesthesia (Nervous system disorders) | 4/180 | 1/176
Sedation (Nervous system disorders) | 7/180 | 7/176
Somnolence (Nervous system disorders) | 15/180 | 6/176
Euphoric mood (Psychiatric disorders) | 4/180 | 0/176
Insomnia (Psychiatric disorders) | 5/180 | 1/176
Cough (Respiratory, thoracic and mediastinal disorders) | 2/180 | 6/176

LIMITATIONS AND CAVEATS:
Further enrollment in this study was stopped based on the recommendation of an independent Data Monitoring Committee (DMC). An interim data analysis did not suggest the potential for robust efficacy. The study was not stopped for any safety findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.